CLINICAL TRIAL: NCT02280655
Title: Adverse Effects of Red Blood Cell Transfusions: A Unifying Hypothesis
Brief Title: Adverse Effects of Red Blood Cell Transfusions: A Unifying Hypothesis (Aim 3)
Acronym: INOBA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, John D Roback, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00015316a
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Cardiovascular Diseases
Keywords: Blood Transfusions
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Storage-aged red blood cells (saRBCs) (Active Comparator): Subjects with cardiovascular disease (CVD) received a transfusion with older stored red blood cells (RBCs) units. The units had been stored for greater than 21 days.
  Interventions: Biological: Storage-aged red blood cells (saRBCs) units
- Fresh red blood cells (RBCs) (Active Comparator): Subjects with cardiovascular disease (CVD) received a transfusion with fresh red blood cells (RBCs) units. The units had been stored for less than 14 days.
  Interventions: Biological: Fresh red blood cells units

INTERVENTIONS:
Biological: Storage-aged red blood cells (saRBCs) units — Packed RBCs units stored for greater than 21 days, with a mean storage duration of 29.6 ± 4.9 days (mean ± SD)
  Arms: Storage-aged red blood cells (saRBCs)
Biological: Fresh red blood cells units — Packed RBCs units stored for less than 14 days, with a mean storage duration of 9.6 ± 3.9 days (mean ± SD)
  Arms: Fresh red blood cells (RBCs)

SUMMARY:
Transfusion of red blood cells is often used in critically ill patients with low red blood cell counts to prevent disease progression and death. Recent studies suggest that the use of "aged" versus "fresh" red blood cells are associated with worse clinical outcomes. There is evidence that red blood cells work with the cells lining our blood vessels to produce a variety of substances that normally cause arteries to relax and increase blood supply. Two of these substances are called nitric oxide (NO) and endothelium-derived hyperpolarizing factor (EDHF). The investigators are trying to determine the nature of these substances in human beings when they are transfused "aged" versus "fresh" red blood cells. The purpose of the study is to test the effects of transfusing "aged" versus "fresh" red blood cells in volunteers with traditional cardiovascular risk factors (high blood pressure, diabetes, high cholesterol, and tobacco use) on 1) the degree of relaxation in the arteries and subsequent changes in blood flow, 2) blood levels of oxidant molecules, 3) inflammation, and 4) stem cells.

A similar study with healthy volunteers are further described in NCT00838331.

DETAILED DESCRIPTION:
Transfusion of red blood cells (RBCs) is often effective at preventing morbidity and mortality in anemic patients. In contrast, recent studies indicate that some RBC components may have functional defects ("RBC storage lesions") that actually cause morbidity and mortality when transfused. For example, patients transfused with RBCs stored >14 days have statistically worse outcomes than those receiving "fresher" RBC units. In addition to the age of stored RBCs, the volume transfused may be important. The Transfusion Requirements in Critical Care (TRICC) study showed that specific patients whose transfusions were limited by a restrictive trigger (RBCs transfusions only when hemoglobin [Hb] < 7 g/dL) had significantly better outcomes than those transfused with a more liberal trigger ([Hb] < 10 g/dL Hb). This finding has been particularly difficult to understand since conventional wisdom suggests that an elevated [Hb] should be beneficial because it supports increased oxygen (O2) delivery. Recipient-specific factors may also contribute to the occurrence of these adverse events. Unfortunately, these events have been difficult to investigate because up to now they have existed only as "statistical occurrences" of increased morbidity and mortality in large data sets. There are currently no clinical or laboratory methods to detect or study them in individual patients.

The microcirculation is composed of a continuum of small vessels including small arterioles, capillaries, and post-capillary venules. The microcirculation represents an actively-adjusting vascular circuit that matches blood flow (and O2 delivery) to local tissue oxygen demands. While the physiologic mechanisms that match O2 delivery to local requirements are incompletely understood, endothelium-derived nitric oxide (NO) clearly plays an important role. Interestingly, recent work has revealed that in addition to transporting O2 and carbon dioxide (CO2), the RBC also controls local NO concentrations and thus may also play a surprisingly important role in regulating blood flow in the microcirculation.

Herein, the investigators bring together previously unconnected data to propose a unifying hypothesis, centered on insufficient NO bioavailability (INOBA), to explain the increased morbidity and mortality observed in some patients following RBC transfusion. In this model, variables associated with RBC units (storage time; 2,3-diphosphoglycerate (2,3-DPG) concentration) and transfusion recipients (endothelial dysfunction; hematocrit [Hct]) collectively lead to changes in NO levels in vascular beds. Under certain circumstances, these variables are "aligned" such that NO concentrations are markedly reduced, leading to vasoconstriction, decreased local blood flow and insufficient O2 delivery to end organs. Under these circumstances, the likelihood of morbidity and mortality escalates. The INOBA hypothesis is attractive because of its explanatory power and because it leads to a number of readily testable predictions, which will be investigated t determine the effects of transfused RBCs in patients with endothelial dysfunction due to cardiovascular disease. A non-invasive ultrasound assay will be used to test whether patients with cardiovascular disease and endothelial dysfunction (who have intrinsic defects in NO synthesis) are more susceptible to adverse effects from stored/processed RBCs (impaired in NO bioavailability) than fresh RBC units. Vasodilation and tissue oxygenation in response to transfusion will be monitored, and Framingham risk scores and cardiovascular disease biomarkers will be tested as potential predictive factors to identify patients most at risk from adverse effects of RBC transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient or outpatient at Emory University Hospital who's physicians have ordered a transfusion of packed red blood cells (pRBCs) of 1 or more units
* Cardiovascular risk factors (hypercholesterolemia, diabetes, hypertension, and tobacco smoking) or known cardiovascular disease) will be carefully documented for each subject

Cardiac risk factors are defined as follows:

* Hypercholesterolemia: Defined as serum low density lipoprotein cholesterol > 140 mg/dL if not currently on lipid-lowering therapy or > 100 mg/dL if on lipid-lowering therapy
* Diabetes: Defined as having fasting blood glucose sample of > 126 mg/dL or a hemoglobin A1c of > 7% or being treated with diabetes medications such as oral hypoglycemic agents, insulin sensitizing agents, or subcutaneous insulin
* Smoking: active tobacco use, 20 cigarettes per day for the past year
* Hypertension: Blood pressure of > 140/90 or currently on anti-hypertensive medications
* Cardiovascular disease: known coronary artery disease by angiogram or documented myocardial infarction

Exclusion Criteria:

* Pregnancy
* Previous transfusion within one week.
* Inability to give informed consent
* On oral or IV nitrate therapy
* On vasopressor agents
* Active illicit drug use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-04; Primary Completion 2012-11 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Roback, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from Emory University Hospital. 142 patients were screened and of those, 99 failed screening or were excluded.
Period: Overall Study
Arm/Group | Storage-aged Red Blood Cells (saRBCs) | Fresh Red Blood Cells (RBCs)
Started | 25 | 18
Completed | 25 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Storage-aged Red Blood Cells (saRBCs) | Fresh Red Blood Cells (RBCs) | Total
Number analyzed (Participants) | 25 | 18 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12) | 60 (15) | 59 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 13 | 11 | 24
Region of Enrollment [Number; unit: participants]
  United States | 25 | 18 | 43

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Flow-mediated Dilation (FMD) After Fresh Red Blood Cells (RBCs) Transfusions vs. Storage-aged Red Blood Cells (saRBCs) Transfusions at Baseline
Description: Ultrasonography of the brachial artery performed at the bedside using a high-resolution 10-megahertz (MHz) ultrasound transducer before and after suprasystolic inflation of a blood pressure cuff for 5 minutes in the ipsilateral upper arm. Brachial artery FMD was calculated as (hyperemic diameter - baseline diameter)/baseline diameter × 100.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of brachial artery diameter
Arm/Group | Storage-aged Red Blood Cells (saRBCs) | Fresh Red Blood Cells (RBCs)
Number analyzed (Participants) | 25 | 18
percentage of brachial artery diameter | 4.87 (5.011) | 5.38 (6.5)

2. Primary Outcome: Brachial Artery Flow-mediated Dilation (FMD) After Fresh Red Blood Cells (RBCs) Transfusions vs. Storage-aged Red Blood Cells (saRBCs) Transfusions at 24 Hours After Transfusion
Description: Ultrasonography of the brachial artery performed at the bedside using a high-resolution 10-megahertz (MHz) ultrasound transducer before and after suprasystolic inflation of a blood pressure cuff for 5 minutes in the ipsilateral upper arm. Brachial artery FMD was calculated as (hyperemic diameter -24 hour diameter)/24 hour diameter × 100.
Time Frame: 24 hours after transfusion
Measure: Mean (Standard Deviation); unit: percentage of brachial artery diameter
Arm/Group | Storage-aged Red Blood Cells (saRBCs) | Fresh Red Blood Cells (RBCs)
Number analyzed (Participants) | 25 | 18
percentage of brachial artery diameter | 2.47 (4.88) | 4.7 (6.19)

ADVERSE EVENTS:
Arm/Group | Storage-aged Red Blood Cells (saRBCs) | Fresh Red Blood Cells (RBCs)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/18
Other Adverse Events (participants affected / at risk) | 0/25 | 0/18

LIMITATIONS AND CAVEATS:
Only patients receiving routine transfusions were included in the study, thus excluding critically ill/actively bleeding patients requiring emergent transfusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes